CLINICAL TRIAL: NCT01625546
Title: Whole Body Hyperthermia and Major Depression (MDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Dr. med. h.c. Erwin Braun Foundation (Unknown); The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other); Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Charles (Chuck) Raison, Clinical Research Professor of Psychiatry, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0147-01
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Whole Body Hyperthermia
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity whole-body infrared heating (Experimental): Subjects will be induced to levels of heat that increases core body temperature to approximately 37.5-38.5 °C using the Whole Body Hyperthermia system.
  Interventions: Device: Whole Body Hyperthermia system
- Low intensity whole-body infrared heating (Sham Comparator): Subjects will be induced to levels of heat that causes only a minor increase in body temperature using Whole Body Hyperthermia system.
  Interventions: Device: Whole Body Hyperthermia system

INTERVENTIONS:
Device: Whole Body Hyperthermia system — The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation. The rise in the body's core temperature is correspondingly rapid and well-tolerated. There are two phases of the thermal challenge, 1) Irradiation phase during which the patient lies recumbent with his/her head positioned outside the tent. The wIRA irradiators are arranged above the exposed upper part of the body; and 2) Heat retention phase during which the patient lies in the chamber with the walls of the tent positioned to retain heat.

SUMMARY:
Major depressive disorder (MDD) is predicted to be the second leading cause of disability worldwide by the year 2020. The economic burden of depression in the United States is significant: $83.1 billion in 2000 and increasing. Much of this burden comes from the high rate of sub-optimal treatment outcomes associated with the disorder. Indeed, only 50% of MDD patients recover in less than 12 weeks with adequate treatment, and up to 20% of patients will fail to adequately respond to all currently available interventions. Moreover, current treatments come at the cost of significant central nervous system (CNS) side effects, further highlighting the need for more effective treatments with fewer side effects. This study will compare temperature ranges from the investigators preliminary studies involving thermoafferent pathways resulting in antidepressant actions with lower temperature ranges not expected to activate these pathways as a control condition, with the goal to evaluate whether previous observations were related to the temperature range in question or can be achieved with other levels.

DETAILED DESCRIPTION:
We will conduct a placebo controlled clinical trial to determine if Whole Body Hyperthermia has antidepressant effects in medically healthy patients with moderate to severe MDD. We plan to recruit a sample of 30 medically healthy individuals with MDD who will be randomized to examine whether WBH will demonstrate an antidepressant effect when compared to a control-WBH condition that will be comprised of very mild heating in the WBH machine (Heckel HT3000). To determine acute and sustained effects of WBH on depression severity, the study will include basic clinical and psychiatric assessments 5 days before and after WBH and follow-up assessments at 2, 4, and 6 weeks following WBH. Additionally, assessments will be conducted during the optional open treatment, 1 week following the open treatment, and at the 3 month follow up. To assess whether WBH affects how individuals relate to other people in their environment, as well as how they spend their time in general and to assess social processes, the study will employ the Electronically Activated Recorder (EAR). Participants will wear the EAR device during the day, while going about their lives over the weekend. This weekend monitoring also includes an actigraphy assessment during which participants will wear an actigraphy device during their waking and sleeping hours. In addition, blood will be obtained at multiple time points to assess plasma concentrations of biological predictors or response and mechanism of action for WBH. This study challenges the existing paradigm by determining if peripheral afferent sensory pathways can be accessed to treat MDD and thus avoid problems of exposing all of the brain to non-selective drugs.

ELIGIBILITY:
Inclusion Criteria for MDD patients:

1. Male or female outpatients aged 18-65.
2. Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
3. In the investigator's opinion, has met DSM-IV-TR criteria for Major Depressive Disorder for at least 4 weeks prior to signing consent, single or recurrent episode, without psychotic features, as the subject's primary psychiatric disorder.
4. Able to communicate in English with study personnel.
5. Has a Hamilton Depression Rating Scale (HDRS) score ≥18 at screening and ≥14 on intervention day.
6. For women of child-bearing potential (i.e., one who is biologically capable of becoming pregnant), must be willing to use a medically acceptable form of birth control or practice abstinence for the duration of her participation in the trial.

Exclusion Criteria for MDD patients:

1. Symptoms of depression which, in the investigator's opinion, are better accounted for by a diagnosis other than Major Depressive Disorder.
2. Any of the following diagnoses, as identified by the psychiatric evaluation or study assessments:

   * A current DSM-IV-TR Axis I diagnosis of Dementia; or
   * Any current DSM-IV-TR Axis II diagnosis (i.e. personality disorder) that would suggest potential noncompliance with the protocol; or
   * A lifetime history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder Type 1; or
   * A diagnosis claustrophobia severe enough that it would impair ability to be in the Heckel HT3000 hyperthermia device
   * A current (or within 12 months prior to the Screening visit) diagnosis of Anorexia Nervosa or Bulimia Nervosa
3. Subject has met DSM-IV criteria for Substance Abuse in the 3 months prior to screening visit, or non-remitted Substance Dependence in the 6 months prior to screening visit.
4. A diagnosis of an anxiety disorder that is considered by the investigator to be of greater source of distress or functional impairment than the patient's depressive symptoms. Subjects with comorbid anxiety disorders not excluded above and considered to be of secondary importance will be permitted in the study.
5. Participation in concurrent formal psychotherapy during the trial, or in the 2 weeks prior to the screening visit.
6. Individuals with a history of having difficulty swallowing food or large capsules will be excluded from participating in the assessment of core body temperature (because swallowing a large sensor pill is required). The ingestible temperature capsules will not be used in subjects with any known or suspected obstructive disease of the gastrointestinal tract including, but not limited to esophageal stricture, diverticulosis and inflammatory bowel disease (IBD), peptic ulcer disease, Crohn's disease, ulcerative colitis; previous gastrointestinal surgery.
7. Subject has a medical condition or disorder that:

   * Is unstable and clinically significant, or:
   * Could interfere with the accurate assessment of safety or efficacy of treatment, including:

     1. individuals who are using prescription drugs that may impair thermoregulatory cooling, including diuretics, barbiturates, and beta-blockers, or antihistamines,
     2. individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
     3. individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
     4. hemophiliacs/individuals prone to bleeding,
     5. individuals with a fever the day of study intervention,
     6. individuals with hypersensitivity to heat,
     7. individuals with recent acute joint injury,
     8. individuals with enclosed infections, be they dental, in joints, or in any other tissues.
8. Clinically significant, in the investigator's opinion, abnormal findings on screening laboratory tests or physical exam.
9. Presence of clinically significant suicide risk, based on the investigator's opinion, or a Columbia Suicide Severity Risk Scale (C-SSRS) suicidal ideation score of 4 or 5. Any suicide attempt within 3 months of the Screening visit is exclusionary.
10. Use of any psychotropic medications for 2 weeks (8 weeks for fluoxetine) prior to initiation of the study, with the exception of hypnotic medications (zolpidem, zaleplon, eszopiclone).
11. Need for any non-protocol psychotropic medication during the trial, with the exception of hypnotics used up to four nights per week.
12. Use of any psychoactive dietary or herbal products in the 2 weeks prior to screening visit 2, or at any time during the trial.
13. Women who are pregnant (HCG pregnancy test at screening, or lactating, or who plan to become pregnant during the study.
14. Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial for depression, as well as drug trials with agents that might affect mood or regulation of body temperature.
15. Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
16. Obesity and overall size of subject. It will be up to the PI's discretion will consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
17. History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
18. History of a cerebral vascular accident
19. History of stroke, epilepsy or cerebral aneurisms
20. Cancer in the last five years.
21. Diabetes mellitus types I or II
22. Any clinically significant autoimmune disease (compensated hypothyroidism allowed)
23. Active alcohol or drug abuse/dependence in the 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HAM-D; derived from the 31-item instrument) | Screening, at intervention, and at weeks 1, 2, 4 and 6 following the intervention. Additionally, at the open treatment, 1 week following the open treatment and at the 3-month follow up.
  To determine acute and sustained effects of Whole Body Hyperthermia (WBH) on depression severity.

SECONDARY OUTCOMES:
Change in QIDS (Quick Inventory of Depressive Symptoms) Score from baseline response | Screening, at intervention, and at weeks 1, 2, 4 and 6 following the intervention. Additionally, at the open treatment, 1 week following the open treatment and at the 3-month follow up.
Core body temperature monitoring | 3 days (over the weekend) at baseline, week 1 and week 4.
  Body temperature will be measured with a Vitalsense unit (Minimitter Respironics, Bend OR). The Vitalsense system includes easy to swallow telemetric capsules about the size of a multivitamin (dimensions 23 cm x 8.7 mm) made of medical grade plastic (biocompatible polycarbonate). After ingestion, pills normally pass between 1 to 5 days (mean 2 ± 1.5 days) and then are discarded. A second pill will be ingested if the pill passes during the study visit. Pill temperature sensors transmit data to a small, battery operated, lightweight, user-worn device that may be worn on a belt or placed in a pocket (Dimensions 120 x 90 x 25 mm; weight 200 grams). The devise can collect up to 10 channels for 240 h without battery replacement or download.
Skin conductance level | On the day of the WBH or control treatment, and at one and 4 weeks following the control/intervention.
  Thermoregulatory cooling will be assessed by 1) skin conductance level (SCL) following the protocol outlined by Ward et al
Heart Rate Variability | On the day of the WBH or control treatment, and at one and 4 weeks following the control/intervention.
  Heart Rate Variability (HRV) will be assessed during the period of SCL collection and will be calculated using both time and frequency domain methodologies.
EAR Assessment | 3 days (over the weekend) at baseline, week 1 and week 4.
  To assess whether WBH affects how individuals relate to other people in their environment, as well as how they spend their time in general and to assess social processes, the study will employ the Electronically Activated Recorder (EAR).
Sleep assessment | 3 days (over the weekend) at baseline, week 1 and week 4.
  To assess how the WBH affects sleep, participants will be given an actigraph to wear on their non-dominant wrist over three days and nights during the weekend assessments at baseline, post-intervention week 1 and study week 4. They will also be instructed to complete a daily sleep diary during the time they wear the sleep watch.
Plasma Concentrations of Biological Predictors of Response and Mechanism of Action for WBH. | Prior to WBH or control, following WBH or control, and at Week 1 and Week 4 follow-up visits.
  Blood samples will be analyzed for physiological measures expected to be impacted by WBH including RNA expression, plasma concentrations of BDNF, and pro- and anti-inflammatory cytokines.
QIDS = Quick Inventory of Depressive Symptoms | Screening, baseline, WBH intervention day, once during the three days following the intervention, and at Week 1, 2, 4 and 6 following intervention. Additionally at the open treatment, 1 week following the open treatment and at the 3-month follow up.
  To determine effects of Whole Body Hyperthermia (WBH) on depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Raison, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Background] Hanusch KU, Janssen CH, Billheimer D, Jenkins I, Spurgeon E, Lowry CA, Raison CL. Whole-body hyperthermia for the treatment of major depression: associations with thermoregulatory cooling. Am J Psychiatry. 2013 Jul;170(7):802-4. doi: 10.1176/appi.ajp.2013.12111395. No abstract available. PMID 23820835
- [Derived] Janssen CW, Lowry CA, Mehl MR, Allen JJ, Kelly KL, Gartner DE, Medrano A, Begay TK, Rentscher K, White JJ, Fridman A, Roberts LJ, Robbins ML, Hanusch KU, Cole SP, Raison CL. Whole-Body Hyperthermia for the Treatment of Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Aug 1;73(8):789-95. doi: 10.1001/jamapsychiatry.2016.1031. PMID 27172277